CLINICAL TRIAL: NCT00828685
Title: Early Functional Outcomes After Closed Reduction Percutaneous Pinning vs. Open Reduction Internal Fixation of Distal Radius Fractures: A Prospective Randomized Trial
Brief Title: Early Functional Outcomes After Closed Reduction With Pinning Versus Open Reduction Internal Fixation of Wrist Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Tamara Rozental, Associate Professor of Orthopedic Surgery, Beth Israel Deaconess Medical Center
Other Study IDs: 2005P000301
Record Dates: First submitted 2009-01-13; First posted 2009-01-26 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Wrist Fractures
Keywords: Return to Work; CRPP; ORIF; Distal Radius
MeSH Terms: conditions — Wrist Fractures

ARMS (2):
- Operative (CRPP) (Active Comparator): If indicated, the wrist fracture would be treated with surgery-the specific operative procedure would be randomized.
  Interventions: Procedure: CRPP
- Operative (ORIF) (Active Comparator): If indicated, the wrist fracture would be treated with surgery-the specific operative procedure would be randomized
  Interventions: Procedure: ORIF

INTERVENTIONS:
Procedure: CRPP — Closed reduction, percutaneous pinning
  Arms: Operative (CRPP)
Procedure: ORIF — Open reduction, internal fixation
  Arms: Operative (ORIF)

SUMMARY:
The purpose of this study is to compare early return to function in patients treated with closed reduction percutaneous pinning and open reduction internal fixation in displaced fractures of the distal radius.

Hypothesis: Wrist range of motion, grip strength and outcome at 2-3 months after injury are better in patients treated with open reduction, internal fixation (ORIF) than in patients treated with closed reduction percutaneous pinning techniques (CRPP). In addition patients treated with ORIF return to work at faster rates.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or greater
* Patient functions independently
* Dorsally displaced, extra-articular fracture (Colles' fracture); or simple intra-articular fracture with a single split between the scaphoid and lunate facets.
* Isolated injury (no other injuries).
* One of the following criteria:

Substantial initial displacement

* Greater than 20 degrees dorsal angulation of the articular surface on the lateral view.
* Greater than 100% loss of apposition.
* Greater than 5 millimeters of shortening by ulnar variance on the posteroanterior radiograph.
* Greater than 2 millimeters articular incongruity (step or gap).
* Both dorsal and volar comminution. Inadequate initial manipulative reduction
* Greater than 5 degrees of dorsal angulation of the articular surface on the lateral radiograph.
* Greater than 3 millimeters of radial shortening by ulnar variance on the posteroanterior radiograph.
* Greater than 2 millimeters articular incongruity.
* Bayonett apposition of the volar cortex.
* Less than 15 degrees of ulnarward inclination of the articular surface in the posteroanterior radiograph. Loss of reduction within 3 weeks of injury.
* Any of the following changes in alignment from the initial post- reduction radiographs qualify:

  * 5 degrees or greater loss of palmar tilt of the articular surface on the lateral radiograph.
  * 2 millimeters or greater loss of radial height by ulnar variance on the posteroanterior radiograph.
  * 5 degrees or greater loss of ulnarward inclination of the articular surface of the distal radius on the posteroanteriorradiograph.
  * 2 millimeters or greater articular incongruity.

Exclusion Criteria:

* More complex articular fractures (i.e. anything more than a simple sagittal split between the scaphoid and lunate facets).
* Volarly displaced fractures.
* Infirm patients.
* Patients that rely on others for basic functional activities.
* Open fractures
* Fractures associated with neurovascular injury.
* Fractures associated with major head, neurological, or visceral injuries that will inhibit the ability to participate in a structured exercise program.
* Associated musculoskeletal injuries to the same arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Wrist range of motion measurement. As well as recorded score from the DASH questionnaire. | 3 months post surgery

SECONDARY OUTCOMES:
Range of motion measured in wrist and a scored DASH questionnaire | 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tamara D Rozental, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Rozental TD, Blazar PE, Franko OI, Chacko AT, Earp BE, Day CS. Functional outcomes for unstable distal radial fractures treated with open reduction and internal fixation or closed reduction and percutaneous fixation. A prospective randomized trial. J Bone Joint Surg Am. 2009 Aug;91(8):1837-46. doi: 10.2106/JBJS.H.01478. PMID 19651939